CLINICAL TRIAL: NCT01239407
Title: Culturally Focused Psychiatric Consultation Service for Asian American and Latino American Primary Care Patients With Depression
Brief Title: Culturally-focused Consultation for Asian Americans and Latino Americans
Acronym: CFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Nhi-Ha T. Trinh, Staff psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-P-000954
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2012-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as usual (No Intervention): The treatment as usual arm consists of two phone or in-person interviews:
  1. Patients are asked questions about their mental health, their views of mental health, and how they cope with their mental health (including any treatment they might be receiving).
  2. Patients are asked the same questions 6 months after the initial interview.
- Culturally focused psychiatric consultation (Experimental): The consultation is comprised of 3 visits:
  1a. Psychiatric diagnostic interview, self-rated questionnaires (in-person consultation).
  1b. Intervention focused on learning about depression and how to treat it using culturally relevant resources.
  2. Follow-up visit two weeks later to go over patients' questions, homework if applicable, and patients' ability to meet the goals outlined in the first visit (in-person or phone visit).
  3. 6-month follow up: 6 months after the initial consultation, patients are asked about mental health symptoms and mental health treatment they might be receiving (phone visit unless patient requests in-person).
  Interventions: Behavioral: Culturally focused psychiatric consultation

INTERVENTIONS:
Behavioral: Culturally focused psychiatric consultation — The consultation is comprised of 3 visits:
  1a. Psychiatric diagnostic interview, self-rated questionnaires (in-person consultation).
  1b. Intervention focused on learning about depression and how to treat it using culturally relevant resources.
  2. Follow-up visit two weeks later to go over patients' questions, homework if applicable, and patients' ability to meet the goals outlined in the first visit (in-person or phone visit).
  3. 6-month follow up: 6 months after the initial consultation, patients are asked about mental health symptoms and mental health treatment they might be receiving (phone visit unless patient requests in-person).
  Arms: Culturally focused psychiatric consultation

SUMMARY:
The purpose of this study is to determine if a culturally focused psychiatric (CFP) consultation service can improve depressive symptoms and increase diagnosis and treatment of depression in Asian American and Latino American primary care patients at the Massachusetts General Hospital.

DETAILED DESCRIPTION:
This study's aim is to determine if a culturally focused mental health consultation will help Latino and Asian Americans who are experiencing sadness, stress, or other symptoms of depression. Eligible adults must already have a primary care physician at Massachusetts General Hospital.

In this study, patients will be randomly assigned, like the flip of a coin, to receive the culturally focused intervention or treatment as usual. Those who receive the intervention will have three sessions with study personnel, during which they will generally discuss and learn techniques for dealing with their mental health. Those who receive treatment as usual, meaning the regular care they receive through their primary care practice, will have two sessions with study personnel during which they will generally discuss their mental health. All study visits and patient materials are provided in patients' language of choice - English, Spanish, Mandarin, Cantonese, or Vietnamese. All patients will be compensated for completing study visits.

About half of the study patients in both arms will also be invited to participate in optional qualitative interviews, in which they will be asked questions about their expectations for the research study and their ideas for improving culturally sensitive mental health services. In addition, a small sample of Asian American patients who did not participate in the study but who have PCPs at the sites where the study was conducted will be contacted for a qualitative interview. This interview will address reasons why Asian American recruitment for the study was so challenging.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent
* Adults 18 years of age or older
* Members of either Asian American or Latino American minority groups
* Currently experiencing depressive symptoms

Exclusion Criteria:

* Active unstable, untreated psychiatric illness precluding participation in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To determine if a culturally focused psychiatric (CFP) consultation service can improve depressive symptoms and increase diagnosis and treatment of depression in Asian American and Latino American primary care patients at MGH. | 6 months after baseline assessment

SECONDARY OUTCOMES:
To determine the feasibility and cost associated with implementing a CFP consultation service within a primary care setting at MGH. | Two years after study enrollment began

CONTACTS AND LOCATIONS:
Overall Officials: Nhi-Ha Trinh, M.D., MPH, Principal Investigator — Massachusetts General Hospital; Andres Bedoya, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kirmayer LJ, Thombs BD, Jurcik T, Jarvis GE, Guzder J. Use of an expanded version of the DSM-IV outline for cultural formulation on a cultural consultation service. Psychiatr Serv. 2008 Jun;59(6):683-6. doi: 10.1176/ps.2008.59.6.683. PMID 18511590
- [Background] Yeung A, Yu SC, Fung F, Vorono S, Fava M. Recognizing and engaging depressed Chinese Americans in treatment in a primary care setting. Int J Geriatr Psychiatry. 2006 Sep;21(9):819-23. doi: 10.1002/gps.1566. PMID 16955440
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Derived] Trinh NH, Bedoya CA, Chang TE, Flaherty K, Fava M, Yeung A. A study of a culturally focused psychiatric consultation service for Asian American and Latino American primary care patients with depression. BMC Psychiatry. 2011 Oct 13;11:166. doi: 10.1186/1471-244X-11-166. PMID 21995514